CLINICAL TRIAL: NCT06074354
Title: Assessing the Use of MY-RIDE, a Just-in-time Adaptive Intervention, to Improve HIV Prevention and Substance Use in Youth Experiencing Homelessness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Diane Santa Maria, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SN-23-0360; 1R01NR020997-01A1 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-10-10 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MY-RIDE group (Experimental)
  Interventions: Behavioral: MY-RIDE group
- Attention-control group (Active Comparator)
  Interventions: Behavioral: Attention-control group

INTERVENTIONS:
Behavioral: Attention-control group — Participants will receive a one-hour general health promotion session from a nurse and be issued a phone that will deploy the EMA on the same schedule as the intervention arm. They will also receive usual care from the clinics, drop-in center, and shelter recruitment sites. Usual care includes accessing social workers and case managers for immediate housing, food, and clothing needs and assistance in navigating the local Continuum of Care system to access social services.
  Arms: Attention-control group
Behavioral: MY-RIDE group — MY-RIDE has three main components: 1) One nurse-led face-to-face session; 2) three months of Ecological Momentary Assessments (EMA) with personalized messaging delivered by phone in real-time in response to one's current risk; and 3) access to on-demand healthcare/PrEP navigation and referrals.
  Arms: MY-RIDE group

SUMMARY:
The purpose of this study is to determine whether Motivating Youth to Reduce Infections, Disconnections, and Emotion dysregulation (MY-RIDE) decreases substance use , to determine whether MY-RIDE increases human immunodeficiency virus (HIV) prevention strategies and to evaluate MY-RIDE effects on willingness to take Pre-Exposure Prophylaxis (PrEP), stress, substance use urge, and use of mental health and substance use services when compared to attention control youth

ELIGIBILITY:
Inclusion Criteria:

* have engaged in substance use (alcohol or illicit drugs)
* speak English
* are experiencing homelessness
* engaged in sexual activity in the last 6 months or plan to in the next month
* are not planning to move out of the metro area during the 15-month study period.

Exclusion Criteria:

* Youth Experiencing Homelessness (YEH) who have low literacy based on the Rapid Estimate of Adult Literacy in Medicine-Short Form (scores < 4)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in substance use | baseline, end of intervention (3 months after baseline), 3 months after intervention, 6 months after intervention, and 12 months after intervention

SECONDARY OUTCOMES:
Change in condom use | baseline, end of intervention (3 months after baseline), 3 months after intervention, 6 months after intervention, and 12 months after intervention
Change in PrEP uptake as assessed by the self reported tool | baseline, end of intervention (3 months after baseline), 3 months after intervention, 6 months after intervention, and 12 months after intervention
  PrEP uptake is defined as the self initiation of HIV prevention medication
Change in sexually transmitted infections (STIs) | baseline, end of intervention (3 months after baseline), 3 months after intervention, 6 months after intervention, and 12 months after intervention
  This will be assessed by a blood test to detect biomarkers for HIV and Syphilis, and urine test for Gonorrhea and Chlamydia

CONTACTS AND LOCATIONS:
Overall Officials: Diane M Santa Maria, DrPH, MSN, RN, PHNA-BC, FSAHM, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santa Maria D, Padhye N, Businelle M, Slesnick N, Ricondo S, Lightfoot M. Just-in-Time Adaptive Intervention to Improve HIV Prevention and Substance Use in Youth Experiencing Homelessness (MY-RIDE): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Oct 10;14:e78006. doi: 10.2196/78006. PMID 41072013